CLINICAL TRIAL: NCT04940234
Title: Patient Perceptions of Physician Education and Quality by Race
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Marcella Alsan, Principal Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB21-0682
Record Dates: First submitted 2021-06-07; First posted 2021-06-25 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Racism; Bias, Racial
Keywords: healthcare
MeSH Terms: conditions — Racism

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Black Expert (Experimental): Survey respondents are exposed to a Black person wearing expert attire.
  Interventions: Behavioral: Exposure to a Photo
- Black Layperson (Experimental): Survey respondents are exposed to a Black person wearing layperson's attire.
  Interventions: Behavioral: Exposure to a Photo
- White Expert (Experimental): Survey respondents are exposed to a white person wearing expert attire.
  Interventions: Behavioral: Exposure to a Photo
- White Layperson (Experimental): Survey respondents are exposed to a white person wearing layperson's attire.
  Interventions: Behavioral: Exposure to a Photo

INTERVENTIONS:
Behavioral: Exposure to a Photo — We plan to recruit subjects and randomly assign them to one of four treatments. In each treatment arm, the subject will view a photo of a man. We experimentally vary treatment along two dimensions: whether the man is wearing expert vs. layperson attire and whether the man is white vs. black. We will survey participants' beliefs about the actors' educational attainment and perceived quality as measured by subjects' willingness to accept medical advice for non-urgent health issues or participate in a clinical trial being led by the individual in the photo.

SUMMARY:
Research has documented positive effects of doctor-patient race concordance, suggesting that increasing diversity among healthcare professionals may play an important role in addressing well-documented racial health disparities in the US. It also remains critical to improve the quality of interactions in race discordant doctor-patient relationships. However, as health systems consider policies to increase the number of minority healthcare professionals, especially among doctors, questions about the equilibrium effects of such initiatives naturally emerge. In this project, the investigators examine whether and how patients vary their perceptions of healthcare professionals by race.

DETAILED DESCRIPTION:
Research has documented positive effects of doctor-patient race concordance. Given the low representation of minorities among doctors in the US, this evidence suggests that the path to addressing well-documented racial health disparities involves both increasing diversity among healthcare professionals and improving the quality of interactions in race-discordant doctor-patient relationships. Increased focus on improving minority representation among healthcare professionals, and especially among doctors, naturally raises questions about the equilibrium effects of such initiatives. In this study, the investigators aim to explore one potential avenue for equilibrium effects. A growing literature examines how doctors' behavior and beliefs change with patient race and potentially affect the quality of healthcare interactions. This project examines whether and how patients vary their perceptions of the quality of doctors based on race. Significant variation in the perceived quality of minority healthcare professionals could adversely affect the quality and effectiveness of healthcare interactions involving these professionals. Moreover, the range of potential negative patient attitudes that could be encountered in day-to-day clinical practice may also be considered an anticipatory tax and another barrier for prospective minority trainees.

This projects aim to test the following hypotheses: (1) whether subjects believe Black experts are less educated compared with White experts; (2) whether subject believe Black experts are lower quality compared with White experts; (3) whether there is any variation in these two outcomes based on respondent race. The investigators also explore a potential mechanism by examining the extent to which differences in patients' beliefs about the likely occupation of individuals explains differences in patients' beliefs about educational attainment and quality. In this case, the investigators hypothesize that the race of the individual in the photo may be affecting the weight that individuals put on the "expert attire" treatment.

ELIGIBILITY:
Inclusion Criteria:

- participant identifies as Black or White

Exclusion Criteria:

* participant doesn't identify as Black or White
* younger than 25 years old

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Willingness to Accept Medical Advice | 6 months
  Survey respondents' willingness to accept the medical advice of the man in the photo.
Willingness to Participate in a Clinical Trial | 6 months
  Survey respondents' willingness to participate in a clinical trial led by the man in the photo.
Education Perception | 6 months
  Survey respondents' perceived education of the man in the photo.
Occupation Perception | 6 months
  Survey respondents' perceived occupation of the man in the photo.

SECONDARY OUTCOMES:
Willingness to Wait | 6 months
  Survey respondents' willingness to wait for their preferred healthcare provider.
Perceived Attractiveness | 6 months
  Survey respondents' perceived attractiveness of the man in the photo.

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No